CLINICAL TRIAL: NCT04683653
Title: RT-PACE: Phase I/II Study of Adjuvant Whole Pelvic Hypofractionated Radiotherapy for Non-Metastatic Cervical and Endometrial Cancer
Brief Title: Study of Pelvic Hypofractionated Radiotherapy in Endometrial Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IRB20-1390
Record Dates: First submitted 2020-12-21; First posted 2020-12-24 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Radiation Dose Hypofractionation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hypofractionated Radiation Treatment (Dose-Finding Arm) (Experimental): All study participants in this arm will receive hypofractionated whole pelvic radiation treatment for a shortened time period of 3-5 weeks. The goal of this arm is to establish a safe and tolerable dose of shortened (hypofractionated) pelvic radiation treatment for study participants. Once a safe and tolerable dose is established for this shortened form of radiation treatment, participants who meet criteria for the second phase of this study will participate in an expansion cohort that will explore the efficacy (how effective shortened/hypofractionated radiation treatment is for treating endometrial cancer).
  Interventions: Radiation: Hypofractionated Radiation
- Expansion Cohort (Efficacy Arm) (Experimental): Participants in this arm will test how effective hypofractionated/shortened whole radiation treatment is ("efficacy") at the dose established in the first phase of this study by following up with their doctors to report their current health status and symptoms during clinical visits. Participants will return for routine clinical follow-up approximately 1 month following radiation, then at 3 months following radiation, then every 3 months for the next 2 years following treatment.
  Interventions: Other: Clinical Follow-Up and Assessments

INTERVENTIONS:
Radiation: Hypofractionated Radiation — Radiation treatment in which the total dose of radiation is divided into large doses and treatments are given less often. Hypofractionated radiation therapy is given over a shorter period of time (fewer days or weeks) than standard radiation therapy.
  Arms: Hypofractionated Radiation Treatment (Dose-Finding Arm)
Other: Clinical Follow-Up and Assessments — At each visit, the subject will be evaluated for any signs of their endometrial cancer or symptoms returning (clinical disease recurrence) and any negative side effects associated with their prior radiation treatment. Study participants will also be asked to fill out a survey regarding bowel/urinary habits and quality of life questionnaires (known as the "EPIC questionnaire") during these visits. The data collected during these clinical follow up visits will be used to determine how effective hypofractionated/shortened whole radiation therapy is for treating endometrial cancer.
  Arms: Expansion Cohort (Efficacy Arm)

SUMMARY:
This study will investigate if a shorter treatment course (known as "hypofractionation") for pelvic radiation is safe for women with endometrial cancer. Doctors leading the study will also determine the safest and most tolerable dose of shortened radiation (hypofractionation) used to treat women in this study. Because this study will shorten the radiation course typically used to treat endometrial cancer, each daily treatment given to women in this study will be slightly higher than normal to ensure that the total radiation dose they receive is still effective and similar to the radiation dose they would receive if they were not participating in this study (standard treatment).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary cervical cancer or uterine cancer of any histology
* Age ≥ 18 years.
* Non-metastatic disease according to the International Federation of Gynecology and Obstetrics (FIGO).
* Must have been treated with definitive intent, including standard-of-care hysterectomy, without any gross residual disease post-operatively. Nodal dissection is not required, but if it is not performed, then diagnostic imaging to confirm absence of gross pelvic or para-aortic disease should be obtained pre- or post-operatively.
* Recommended to undergo whole pelvic radiotherapy without concurrent chemotherapy or para-aortic radiation. Chemotherapy before or after radiotherapy is acceptable.
* Eastern Cooperative Oncology Group (ECOG) PS≤ 2
* Able to provide informed consent and willingness to sign an approved consent form

Exclusion Criteria:

* Distant metastases as determined clinically or radiographically based upon standard-of-care work-up for endometrial cancer.
* Concurrent (or other) chemotherapy occurring at the time of study.
* Gross residual disease (cancer cells that remain after attempts to remove the cancer have been made) post-operatively and/or at the time of radiation based upon pre-op or post-op imaging, intra-operative findings, and gynecologic oncologists' judgment.
* History of small bowel obstruction, inflammatory bowel disease, irritable bowel syndrome, connective tissue disorder requiring ongoing active medical management, or prior radiation therapy directed to the pelvis.
* Unresolved grade 2 or higher chemotherapy-associated diarrhea or abdominopelvic pain requiring medication prior to the initiation of radiation.
* Recommendation to undergo para-aortic nodal irradiation.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 100 (Estimated)
Dates: Start 2021-01-15 (Actual); Primary Completion 2027-05-22 (Estimated); Study Completion 2027-05-22 (Estimated)

PRIMARY OUTCOMES:
The Maximum Tolerated Dose of Hypofractionated Whole Pelvic Radiation Treatment (Phase 1) | 3-5 weeks
  The maximum tolerated dose-per-fraction regimen of whole pelvic radiation therapy that will be administered during uterine cancer treatment.
Change in patient-reported acute gastrointestinal side effects after completion of hypofractionated radiation (Phase 2) | 3-5 weeks (end of treament)
  Change in quality-of-life experience on the bowel and urinary domains

SECONDARY OUTCOMES:
Change in patient-reported acute urinary side effects | 1 month post radiation
  Determined using frequency of reported events of urinary frequency, urinary incontinence, and urinary urgency on the Patient Reported Outcomes (PRO-CTCAE)
Change in gastrointestinal toxicity over time | 1 month post radiation
  Determined using frequency of reported events of diarrhea and proctitis on the Patient Reported Outcomes (PRO-CTCAE)
Overall quality of life after treatment | 2 years post treatment
  Total quality of life score from the Functional Assessment of Cancer Therapy (FACT)-General questionnaire will be calculated. A higher score indicates better quality of life.
Financial Distress of Treatment | End of treatment
  Change in reported financial distress in patients as reported on the Functional Assessment of Chronic Illness Therapy- COST (FACIT-COST) questionnaire. Higher scores on scale of 0-5 indicates better financial wellbeing.
Treatment Satisfaction | End of treatment
  We will characterize the measure of regret experienced in the study patients over time as reported on the Decision Regret Scale questionnaire. Higher scores on scale of 0-100 indicates high regret.

CONTACTS AND LOCATIONS:
Overall Officials: Christina Son, MD, Principal Investigator — University of Chicago
Locations (5):
- United States (5):
  - Winship Cancer Institute, Emory University, Atlanta, Georgia
  - University of Illinois at Chicago (UIC), Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - MD Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah